CLINICAL TRIAL: NCT03883542
Title: Sub-type Specific Genomic Mutations in Serous Borderline Ovarian Tumors
Brief Title: Sub-type Specific Genomic Mutations in sBOTs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Stefan Cosyns, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: sBOT
Record Dates: First submitted 2019-02-26; First posted 2019-03-21 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Ovarian Neoplasm Epithelial
Keywords: low malignant potential; serous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Macrodissection of borderline ovarian tumor tissue. DNA extraction from paraffin embedded material for genetic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- serous BOT: simple serous BOT ovarian tissue
  Interventions: Genetic: genomic mutations study
- serous BOT with non-invasive implants: BOT ovarian tissue presenting with non-invasive implants
  Interventions: Genetic: genomic mutations study
- sBOT with micropapillary grow pattern: BOT ovarian tissue presenting with micropapillary grow pattern
  Interventions: Genetic: genomic mutations study
- serous BOT with invasive implants: sBOT ovarian tissue presenting with invasive implants at the time of diagnosis
  Interventions: Genetic: genomic mutations study

INTERVENTIONS:
Genetic: genomic mutations study — Sequencing of the DNA samples extracted from the subgroups
  1. serous BOT tissue,
  2. serous BOT tissue with non-invasive implants and
  3. serous BOT tissue with micropapillary grow pattern will undergo a panel testing for Type 1 genes (small panel 15-40 mutations) AND p53 AND BRCA testing
  Sequencing of the DNA samples extracted from the serous BOT tissue with invasive implants will undergo a more comprehensive examination (large panel +- 1000 genes checked)

SUMMARY:
The aim of this study is to identify different origin in carcinogenesis between serous borderline ovarian tumors presenting a. without implants, b. with non-invasive implants, c. with invasive implants and d. with micropapillary pattern.

The presence of specific mutations could suggest for a more aggressive primary treatment if a higher risk of recurrence can be expected.

DETAILED DESCRIPTION:
Introduction Borderline Ovarian Tumors (BOTs) behave indolently in the vast majority of cases and the prognosis is usually favorable. There is more evidence that two subtypes of BOTs represent a higher risk of recurrence or even progression to an invasive ovarian cancer. In case of a presentation with a micro-papillary grow pattern or when invasive implants are diagnosed the prognosis tend to be less favorable.

Genome sequencing in ovarian cancer helped to differentiate two different pathways in the carcinogenesis.

Low grade serous carcinomas evolving from adenofibromas or borderline tumors over non-invasive micropapillary serous borderline tumors to invasive micropapillary serous carcinoma, show frequent mutations in the Kirsten Rat Sarcoma gene (KRAS), B-Raf Kinase gene(BRAF), Erb-B2 Receptor Tyrosine Kinase 2 gene (ERBB2), Phosphatase and Tensin homolog gene (PTEN), Phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha gene (PIK3CA) and Catenin Beta 1 gene (CTNNB1). This pathway is called Type I and is characterized by a slow step-wise process. These low-grade invasive tumors are indolent and are known with a better outcome than high-grade invasive tumors.

In contrast the Type II pathway development of invasive tumors is rapid and vast majority of tumors show a Tumor Protein p53 (TP53) mutation and loss of Breast Cancer type 1 susceptibility protein (BRCA1).

The aim of this study is to identify different origin in carcinogenesis between serous borderline ovarian tumors presenting a. without implants, b. with non-invasive implants, c. with invasive implants and d. with micropapillary pattern.

The presence of specific mutations could suggest for a more aggressive primary treatment if a higher risk of recurrence can be expected.

ELIGIBILITY:
Inclusion Criteria:

* Paraffin embedded material from the original borderline ovarian tumor must be present and of good quality for DNA extraction.
* Original slides are available for central pathological review.

Exclusion Criteria:

* Presence of invasive ovarian carcinoma.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven serous bordeline ovarian tumors.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
genetic mutations | 2020
  amount and type of genetic mutations in different subgroups will be analyzed and compared between the different subgroups. Are the mutations suggestive for a type I or type II pathway differentiation?

CONTACTS AND LOCATIONS:
Overall Officials: stef cosyns, dr, Principal Investigator — UZBrussel
Locations (1):
- Universitair Ziekenhuis UZBrussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morice P, Uzan C, Fauvet R, Gouy S, Duvillard P, Darai E. Borderline ovarian tumour: pathological diagnostic dilemma and risk factors for invasive or lethal recurrence. Lancet Oncol. 2012 Mar;13(3):e103-15. doi: 10.1016/S1470-2045(11)70288-1. PMID 22381933
- [Background] Vang R, Shih IeM, Kurman RJ. Ovarian low-grade and high-grade serous carcinoma: pathogenesis, clinicopathologic and molecular biologic features, and diagnostic problems. Adv Anat Pathol. 2009 Sep;16(5):267-82. doi: 10.1097/PAP.0b013e3181b4fffa. PMID 19700937
- [Background] Despierre E, Lambrechts D, Neven P, Amant F, Lambrechts S, Vergote I. The molecular genetic basis of ovarian cancer and its roadmap towards a better treatment. Gynecol Oncol. 2010 May;117(2):358-65. doi: 10.1016/j.ygyno.2010.02.012. Epub 2010 Mar 7. PMID 20207398
- [Background] Kurman RJ, Shih IeM. The origin and pathogenesis of epithelial ovarian cancer: a proposed unifying theory. Am J Surg Pathol. 2010 Mar;34(3):433-43. doi: 10.1097/PAS.0b013e3181cf3d79. PMID 20154587